CLINICAL TRIAL: NCT04508127
Title: A Prospective Open Label Feasibility Study to Investigate the Dynamic Brain Imaging in Patients With Intractable Neuropathic Pain Routinely Treated With Targeted Spinal Cord Stimulation
Brief Title: A Feasibility Study to Investigate the Dynamic Brain Imaging in Patients Following SCS- DRG
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 15.LO.1667
Record Dates: First submitted 2019-01-15; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2018-11

CONDITIONS: Neuropathic Pain
Keywords: DRG; SCS; PET Scans
MeSH Terms: conditions — Neuralgia | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Active Procedure: The patients will receive targeted Percutaneous Spinal Cord Stimulation at suitable DRG with Axium SCS system as part of their standard treatment for lumbar pain. The lead placement will happen in 2 stages. First stage involves placement of leads and an externalised device and is a trial stage. Patient deemed to have a good response to first stage will proceed to the second stage to have the permanent implant. Again this is part of our standard care. Normally our drop out rate after first stage is less than 10% and these patients will not have subsequent tests including PET-CT scan and questionnaires.
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation

SUMMARY:
Targeted SCS is a standard and safe interventional pain procedure that is offered to patients with intractable neuropathic pain for their symptomatic relief. The known and reported complications include technical failure to perform the procedure, failure to gain symptomatic relief, trauma to nerve, and infection. These risks are very low in incidence and part of any interventional pain procedure in the spine.

PET-CT scan involves insertion of a cannula and administration of a dye (FDG) as a contrast in a patient who has been fasted for at least 6 hours. The procedure is lengthy and can take up to 2 to 3 hours. This includes a 30-60 minute resting time following the injection of contrast. The actual scan itself takes up to 30 minutes. There is a small chance of pain and redness at the injection site. Allergic reaction to the radio-contrast is rare and is usually mild. Patients with known allergy to FDG will not be recruited in the study. Some patients can feel claustrophobic at the time of the scan which can make them feel anxious. The PET-CT scan involves radiation with associated risks as detailed in the previous section. All these risks will be explained to the patients at the time of the informed consent.

DETAILED DESCRIPTION:
Targeted Spinal Cord Stimulation (SCS) using dorsal root ganglion (DRG) stimulation is an effective therapy for a number of different chronic painful conditions of neuropathic origin. British Pain Society has issued a detailed list of indications for SCS which includes intractable neuropathic of various ethiologies. These patients may present with both peripheral and central sensitisation, clinically manifested as hyperalgesia and allodynia.

The National Institute for Health and Care Excellence (NICE- TA 159) has issued full guidance to the NHS in England, Wales, Scotland and Northern Ireland on SCS for chronic pain of neuropathic or ischemic origin. However much debate still exists about the exact mechanism and the pathways remain to be elucidated.

The neural pathway at the level of Dorsal root ganglion (DRG) is well described in anatomical dissections. DRG is no longer considered a passive anatomical structure but is an important junction in the pain pathway through which both afferent and efferent pain impulses are transmitted and there by the pathway is modulated.

Targeting DRG using both local anaesthetic and steroid as well as radiofrequency are well recognised techniques for managing patients with neuropathic back and leg pain both with and without previous surgery. It is a common practice for patients with radicular type back pain to undergo a trial of intervention such as DRG injection prior to undergoing surgery.

A growing body of evidence is emerging to support the use of targeted SCS at the level of DRG. Targeted SCS is a chronic pain management technique targeting the DRG - a cluster of sensory neurons that serve as a conduit of pain signals from the peripheral nervous system to the central nervous system. By stimulating this structure, pain signals can be blocked before they are transmitted to the spinal cord and processed in the brain. Unlike traditional SCS therapy, which targets nerves along the spinal cord's dorsal column, DRG stimulation offers selective targeting of pain areas, with fewer side effects, such as paresthesias. This will allow us to target more specific dermatomes and there by treating a much larger number of neuropathic pains including more localised lesions. The strongest evidence for the successful use of targeted SCS emerges from the 'ACCURATE' study which is a large a large multicentre study conducted in the United States of America. The ACCURATE study showed that DRG stimulation using the Axium system was better than traditional SCS (81.2 vs 55.7 percent) in providing pain relief. Participants also reported no differences in the intensity of paresthesias due to postural changes, a common side effect of traditional SCS therapy, while using the targeted SCS during the three-month trial. They also reported feeling less stimulated outside their area of pain, demonstrating the precision of DRG stimulation. The results of the U.S. study is also supported by a number of international, peer-reviewed scientific abstracts from Australia and Europe highlighting positive clinical outcomes of targeted SCS for the treatment of chronic, intractable pain.

Dynamic brain imaging is increasingly used as a research tool to understand the mechanisms of pain and also pain interventions. This is done by using either a functional MRI (fMRI) or Positron Emission Tomography (PET-CT). The implant used for neuromodulation for targeted SCS is not MRI compatible which precludes the use of fMRI. Hence PET-CT is the best available option to investigate the changes in the brain in patients having a targeted SCS. Functional changes in the brain are identified by the changes in the regional cerebral blood flow (rCBF) as determined by the changes in the distribution of the radioactiove contrast F18- fluorodeoxyglucose (FDG) in different areas of the brain.

Chronic pain has been associated with changes in brain structure as well as metabolism especially in the second somatic (SII) regions, insula and anterior cingulate cortex (ACC). Less consistently, changes have also been seen in thalamus and primary somatic area (SI). Sensory discrimination, summation, affect, cognition and attention all seem to influence different areas of the brain there by modulate the patient's pain perception. There is some evidence to suggest that some of these changes may be normalised with treatment using either medications or other interventions.

Currently, there is no data looking at the PET-CT scan changes following a targeted SCS. Hence this would be the first study looking into the dynamic brain imaging changes following targeted SCS. This will hopefully give us the information regarding the nature of changes occurring in the brain following a targeted SCS. This will also hopefully enable us to correlate it with the changes inwith QST and health related outcome questionnaires

Patient Preparation and procedure The PET-CT scan will be performed in accordance with the Standard Operating Procedure (SOP) at Barts Health NHS Trust and will be performed at St Bartholomew's hospital. The patient will be fasted for at least 6 hours and the procedure will be explained thoroughly going through all the necessary questions including the IV contrast form if required.

For this procedure, the subject will lie on the table in the PET-CT scanner. At the beginning of each scan, a special contrast called FDG will be injected into an arm vein through a catheter (a thin plastic tube). A special camera records the arrival and disappearance of FDG in various brain areas, creating a picture of the brain's activity in various regions. The required dose of FDG i s is 200 megabecquerel (MBqs) and is given intravenously. The uptake time is 30 minutes from injection to start of the PET-CT scan. The exposure factors of the scanner will be checked and will be set at 120kV (tube voltage) and 50 mAs (tube current). The tube rotation time will be set at 0.5s. The emission time per frame will be set at 3 frames for 5 minutes each.

Following the scan the images will be checked for quality. The 3 dynamic frames will be viewed to check for patient motion and the patient will be discharged if appropriate.

If there is very little (<5mm) motion, the raw data on the PET-CT Recon Server, (PRS) will be reconstructed using the Brain-ctac-suv protocol. The dynamic frames will be summed together. Fused images will be created for storage in the picture archieving and communication system (PACS), the standard system used to store all radiology images in the hospital, archiving, and reporting.

If there is >5mm of motion, it will be reconstructed using the same protocol, but after specifying the time (in seconds) to use best 2 frames if possible. If necessary, 1 frame can be specified. As part of SOP all staff must be trained by an appropriate, qualified staff member to an agreed level of competency and have read and understood this procedure and any other relevant procedures and documentation before they are allowed carry out the procedure.

Safety and radiation dose The FDG-PET Brain scan with a low dose CT for attenuation correction is additional dose due to participation in this study.

The national DRL for an FDG-PET scan for tumour imaging is 250 MBq, giving an effective dose of 5 mSv per scan (ARSAC, 2006). The participating patient will receive a total FDG-PET radiation dose of 16 mSv (from baseline and follow-up scan).

In a patient dose (DLP) audit carried out in March 2015, the low dose Brain CT protocol for PET attenuation correction at St Bartholomew's Hospital gave an effective dose of 0.5 mSv for an average patient (using conversion factors in NRPB-W67, 2005).

The Total Research Protocol Dose in this study is therefore 11 mSv for patients receiving 2 administrations.

The radiation dose from this study therefore falls into risk category III, as defined in ICRP 62 (effective dose > 10 mSv) and is considered a moderate level of risk.

The HPA have endorsed the ICRP recommendation that a nominal risk coefficient of 5 x 10-2 per Sievert is used as the approximate overall fatal risk coefficient (Documents of the HPA, RCE-12, 2009). From this it can be estimated that the lifetime risk of inducing a fatal cancer in a healthy individual from the total research protocol dose is approximately 1 in 1800 for patients receiving 2 administrations. The risk is age dependent and is increased for younger patients, decreasing with age. This should be compared with the natural incidence rate for cancer in the UK.

These factors apply to healthy individuals and should be considered against alleviating the morbidity of the patient's long-term condition.

For comparison, the average annual natural background radiation dose in the UK is 2.2 mSv. The additional radiation dose incurred in this study can be compared to about 5 years' annual background exposure for patients receiving 2 administrations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the age of 18-80 years who has intractable neuropathic pain.
* Minimum baseline pain rating of 50mm on a 100mm NRS in the back and/or leg
* Chronic pain of at least 6 months
* Subject satisfies standard criteria in the study centre for SCS implantation and the NICE 159 criteria for management of intractable neuropathic pain.
* Patients who have given their written informed consent.
* Patient is able and willing to comply with study procedures and follow up schedule.

Exclusion Criteria:

* Female patients of childbearing age who is or plans on becoming pregnant during the course of the study
* Patients who have undergone radiofrequency or injection therapy at or on a target neural structure (DRG) during the past 90 days
* Patient deemed unsuitable to have targeted SCS as assessed by the MDT.
* Patients known to have a condition that in the investigator's judgement precludes participation in the study.
* Patients who have received an investigational drug or have used an investigational device in the 30 days proceeding to study entry
* Patients who are needle phobic or claustrophobic.
* Known allergic reaction to radio-contrast.
* Patients who are at high risk of a radiation hazard (previous radiation induced injury or cancer or previously received high radiation doses).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Pain multi-disciplinary team meetings at Barts Health NHS trust. Patients will be seen by a team of neurosurgeons, pain consultants and psychologist to assess their suitability for targeted SCS.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
The PET-CT and metabolic activity/ mapping at baseline. | baseline
  Determine the presence of a quantifiable alteration in central processing using PET-CT and metabolic activity/ mapping at baseline
The changes of PET-CT and metabolic activity/ mapping at 2 weeks. | 2 weeks
  Determine the presence of a quantifiable alteration in central processing using PET-CT and metabolic activity/ mapping at 2 weeks post treatment.
The changes PET-CT and metabolic activity/ mapping at 4 weeks. | 4 weeks
  Determine the presence of a quantifiable alteration in central processing using PET-CT and metabolic activity/ mapping at 4 weeks post treatment.
The changes PET-CT and metabolic activity/ mapping at 3 months. | 3 months
  Determine the presence of a quantifiable alteration in central processing using PET-CT and metabolic activity/ mapping at 3 months post treatment.
The changes PET-CT and metabolic activity/ mapping at 6 months. | 6 months
  Determine the presence of a quantifiable alteration in central processing using PET-CT and metabolic activity/ mapping at 6 months post treatment.

SECONDARY OUTCOMES:
Pain and satisfaction to treatment assessed using Numerical Rating Scale (NRS) questionnaires at baseline | Baseline
  The changes of SCS on functionality and quality of life in patients before treatment using 11-point NRS scale. The scale is marked 0 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Numerical Rating Scale (NRS) questionnaires at 4 weeks | 4 weeks
  The changes of SCS on functionality and quality of life in patients after treatment using 11-point NRS scale. The scale is marked 0 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Numerical Rating Scale (NRS) questionnaires at 3 months | 3 months
  The changes of SCS on functionality and quality of life in patients after treatment using 11-point NRS scale. The scale is marked 0 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Numerical Rating Scale (NRS) questionnaires at 6 months | 6 months
  The changes of SCS on functionality and quality of life in patients after treatment using 11-point NRS scale. The scale is marked 0 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Numerical Rating Scale (NRS) questionnaires at 12 months | 12 months
  The changes of SCS on functionality and quality of life in patients after treatment using 11-point NRS scale. The scale is marked 0 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Brief Pain Inventory (BPI), questionnaires at baseline | Baseline
  The changes of SCS on functionality and quality of life in patients before treatment BPI questionnaires using a 10 point scale to assess pain, where 1 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Brief Pain Inventory (BPI), questionnaires at 4 weeks | 4 weeks
  The changes of SCS on functionality and quality of life in patients after treatment BPI questionnaires using a 10 point scale to assess pain, where 1 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Brief Pain Inventory (BPI), questionnaires at 3 months | 3 months
  The changes of SCS on functionality and quality of life in patients after treatment BPI questionnaires using a 10 point scale to assess pain, where 1 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Brief Pain Inventory (BPI), questionnaires at 6 months | 6 months
  The changes of SCS on functionality and quality of life in patients after treatment BPI questionnaires using a 10 point scale to assess pain, where 1 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using Brief Pain Inventory (BPI), questionnaires at 12 months | 12 months
  The changes of SCS on functionality and quality of life in patients after treatment BPI questionnaires using a 10 point scale to assess pain, where 1 is no pain and 10 is worst pain.
Pain and satisfaction to treatment assessed using painDETECT at baseline. | Baseline
  The changes of SCS on functionality and quality of life in patients before treatment using Pain DETECT questionnaires. The total score is out of 35 an patients mark their responses to questions which have been marked between 0-5.
Pain and satisfaction to treatment assessed using painDETECT questionnaires at 4 weeks. | 4 weeks
  The changes of SCS on functionality and quality of life in patients after treatment using Pain DETECT questionnaires. The total score is out of 35 an patients mark their responses to questions which have been marked between 0-5.
Pain and satisfaction to treatment assessed using painDETECT questionnaires at 3 months. | 3 months
  The changes of SCS on functionality and quality of life in patients after treatment using Pain DETECT questionnaires. The total score is out of 35 an patients mark their responses to questions which have been marked between 0-5.
Pain and satisfaction to treatment assessed using painDETECT questionnaires at 6 months. | 6 months
  The changes of SCS on functionality and quality of life in patients after treatment using Pain DETECT questionnaires. The total score is out of 35 an patients mark their responses to questions which have been marked between 0-5.
Pain and satisfaction to treatment assessed using painDETECT questionnaires at 12 months. | 12 months
  The changes of SCS on functionality and quality of life in patients after treatment using Pain DETECT questionnaires. The total score is out of 35 an patients mark their responses to questions which have been marked between 0-5.
Pain and satisfaction to treatment assessed using Hospital Anxiety and Depression Scale (HADS) questionnaires at baseline | Baseline
  The changes of SCS on functionality and quality of life in patients before treatment using HADS questionnaires. The questionnaire assesses the depression and anxiety depending on the responses the patient selects for each question. The total questionnaire is scored out of 21 where 11 is maximum for anxiety and 11 is maximum for depression.
Pain and satisfaction to treatment assessed using Hospital Anxiety and Depression Scale (HADS) questionnaires at 4 weeks | 4 weeks
  The changes of SCS on functionality and quality of life in patients after treatment using HADS questionnaires. The questionnaire assesses the depression and anxiety depending on the responses the patient selects for each question. The total questionnaire is scored out of 21 where 11 is maximum for anxiety and 11 is maximum for depression.
Pain and satisfaction to treatment assessed using Hospital Anxiety and Depression Scale (HADS) questionnaires at 3 months | 3 months
  The changes of SCS on functionality and quality of life in patients after treatment using HADS questionnaires. The questionnaire assesses the depression and anxiety depending on the responses the patient selects for each question. The total questionnaire is scored out of 21 where 11 is maximum for anxiety and 11 is maximum for depression.
Pain and satisfaction to treatment assessed using Hospital Anxiety and Depression Scale (HADS) questionnaires at 6 months | 6 months
  The changes of SCS on functionality and quality of life in patients after treatment using HADS questionnaires. The questionnaire assesses the depression and anxiety depending on the responses the patient selects for each question. The total questionnaire is scored out of 21 where 11 is maximum for anxiety and 11 is maximum for depression.
Pain and satisfaction to treatment assessed using Hospital Anxiety and Depression Scale (HADS) questionnaires at 12 months | 12 months
  The changes of SCS on functionality and quality of life in patients after treatment using HADS questionnaires. The questionnaire assesses the depression and anxiety depending on the responses the patient selects for each question. The total questionnaire is scored out of 21 where 11 is maximum for anxiety and 11 is maximum for depression.
Pain and satisfaction to treatment assessed using Pain Self- efficacy Questionnaire (PSEQ) at baseline. | Baseline
  The changes of SCS on functionality and quality of life in patients before treatment using PSEQ questionnaires. Total scores range from 0 - 60 and is done by simple addition. High PSEQ scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.
Pain and satisfaction to treatment assessed using Pain Self- efficacy Questionnaire (PSEQ) at 4 weeks. | 4 weeks
  The changes of SCS on functionality and quality of life in patients after treatment using PSEQ questionnaires. Total scores range from 0 - 60 and is done by simple addition. High PSEQ scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.
Pain and satisfaction to treatment assessed using Pain Self- efficacy Questionnaire (PSEQ) at 3 months. | 3 months
  The changes of SCS on functionality and quality of life in patients after treatment using PSEQ questionnaires. Total scores range from 0 - 60 and is done by simple addition. High PSEQ scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.
Pain and satisfaction to treatment assessed using Pain Self- efficacy Questionnaire (PSEQ) at 6 months. | 6 months
  The changes of SCS on functionality and quality of life in patients after treatment using PSEQ questionnaires. Total scores range from 0 - 60 and is done by simple addition. High PSEQ scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.
Pain and satisfaction to treatment assessed using Pain Self- efficacy Questionnaire (PSEQ) at 12 months. | 12 months
  The changes of SCS on functionality and quality of life in patients after treatment using PSEQ questionnaires. Total scores range from 0 - 60 and is done by simple addition. High PSEQ scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.
Pain and satisfaction to treatment assessed using quality of life EQ5D questionnaires at baseline. | Baseline
  The changes of SCS on functionality and quality of life in patients before treatment using EQ5D questionnaires. An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient. Value nearest to 1 indicate a better quality of life.
Pain and satisfaction to treatment assessed using quality of life EQ5D questionnaires at 4 weeks | 4 weeks
  The changes of SCS on functionality and quality of life in patients after treatment using EQ5D questionnaires. An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient. Value nearest to 1 indicate a better quality of life.
Pain and satisfaction to treatment assessed using quality of life EQ5D questionnaires at 3 months | 3 months
  The changes of SCS on functionality and quality of life in patients after treatment using EQ5D questionnaires. An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient. Value nearest to 1 indicate a better quality of life.
Pain and satisfaction to treatment assessed using quality of life EQ5D questionnaires at 6 months | 6 months
  The changes of SCS on functionality and quality of life in patients after treatment using EQ5D questionnaires. An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient. Value nearest to 1 indicate a better quality of life.
Pain and satisfaction to treatment assessed using quality of life EQ5D questionnaires at 12 months | 12 months
  The changes of SCS on functionality and quality of life in patients after treatment using EQ5D questionnaires. An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient. Value nearest to 1 indicate a better quality of life.